CLINICAL TRIAL: NCT00001300
Title: A Randomized Study of the Effect of Adjuvant Chemotherapy With Doxorubicin and Ifosfamide With Mesna in the Treatment of High-Grade Adult Extremity Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920210; 92-C-0210
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Sarcoma
Keywords: Adjuvant Chemotherapy; Ifosfamide; Randomized Study; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; Mesna

INTERVENTIONS:
Drug: doxorubicin
Drug: ifosfamide
Drug: mesna

SUMMARY:
Randomized study. All patients must be randomized to treatment on Arms I and II within 3 months of definitive surgery on Regimen A.

Regimen A: Surgery followed, as indicated, by Radiotherapy. Amputation; or limb-sparing resection followed by involved-field irradiation using megavoltage equipment with or without electron boost.

Arm I: 2-Drug Combination Chemotherapy with Hematologic Toxicity Attenuation and Urothelial Protection. Doxorubicin, DOX, NSC-123127; Ifosfamide, IFF, NSC-109724; with Granulocyte Colony Stimulating Factor (Amgen), G-CSF,

NSC-614629; and Mesna, NSC-113891.

Arm II: Observation. No adjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients with primary, high-grade soft tissue sarcoma of the extremities will undergo treatment of their primary tumor with either amputation or limb-sparing surgery and radiotherapy, and then be randomized to either observation or adjuvant treatment with doxorubicin and ifosfamide with mesna (with G-CSF) for five cycles beginning post-operatively. Local recurrence, disease-free survival and overall survival will be evaluated in this randomized two-arm trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven AR and ESFT which includes: Classical, atypical and extraosseous Ewing's sarcoma, primitive peripheral neuroectodermal tumors, peripheral neuroepithelioma, primitive sarcoma of bone, and ectomesenchymoma.

Confirmed presence of tumor-specific infusion protein by documented RT-PCR which corresponds to one of the tumor specific peptides available for vaccination.

Measurable tumor.

No prior or current CNS metastases.

PRIOR/CONCURRENT THERAPY:

Arm A patients:

May be enrolled on the protocol for the first phase in the absence of RT PCR documentation of a tumor-specific fusion protein which corresponds to one of the tumor-specific peptides available for vaccination. However, RT PCR documentation at the time of tumor recurrence must occur prior to administration of immunotherapy. At time of initial tumor diagnosis, prior to any cytoreductive therapy.

Arm B patients:

Tumor recurrence occurring during or after receiving at least first line cytoreductive therapy for ESFT and AR. No more than two post-recurrence salvage regimens unless peripheral CD4+T cell number is greater than 400 cells per millimeter cubed.

At least 6 weeks since any treatments and recovered from all acute toxic effects from time in which immunotherapy will be started for this study.

No concurrent estrogen therapy during immunotherapy section of study.

PATIENT CHARACTERISTICS:

Age: 2-25 (at time of initial diagnosis of alveolar rhabdomyosarcoma).

Weight: Greater than 15 kg (at time of apheresis).

Performance status: ECOG 0-2.

Life expectancy: At least 8 weeks.

Hematopoietic:

ANC greater than 100,000/mm3.

Hemoglobin greater than 9.0 g/dL.

Platelet count greater than 50,000/mm3.

Hepatic:

Bilirubin less than 2.0 mg/dL (unless related to involvement by tumor).

Transaminases less than 3 times normal (unless related to involvement by tumor).

Renal:

Creatinine less than 1.5 mg/dL or creatinine clearance greater than 60 mL/min.

Cardiovascular:

No major disorder of cardiovascular system.

Cardiac ejection fraction greater than 40%.

Pulmonary:

No major disorder of pulmonary system.

Other:

Not pregnant or nursing.

HIV negative.

Hepatitis B or C negative.

No patients requiring daily oral corticosteroid therapy.

If allergic to eggs, egg products, or thimerosal, or have a history of Guillain-Barre syndrome, ineligible to receive influenza vaccine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1992-06; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lawrence W Jr, Donegan WL, Natarajan N, Mettlin C, Beart R, Winchester D. Adult soft tissue sarcomas. A pattern of care survey of the American College of Surgeons. Ann Surg. 1987 Apr;205(4):349-59. doi: 10.1097/00000658-198704000-00003. PMID 3566372
- [Background] Alvegard TA, Sigurdsson H, Mouridsen H, Solheim O, Unsgaard B, Ringborg U, Dahl O, Nordentoft AM, Blomqvist C, Rydholm A, et al. Adjuvant chemotherapy with doxorubicin in high-grade soft tissue sarcoma: a randomized trial of the Scandinavian Sarcoma Group. J Clin Oncol. 1989 Oct;7(10):1504-13. doi: 10.1200/JCO.1989.7.10.1504. PMID 2674336
- [Background] Chang AE, Kinsella T, Glatstein E, Baker AR, Sindelar WF, Lotze MT, Danforth DN Jr, Sugarbaker PH, Lack EE, Steinberg SM, et al. Adjuvant chemotherapy for patients with high-grade soft-tissue sarcomas of the extremity. J Clin Oncol. 1988 Sep;6(9):1491-500. doi: 10.1200/JCO.1988.6.9.1491. PMID 3047339